CLINICAL TRIAL: NCT00700583
Title: Alpha-blocker Plus Diuretic Combination Therapy as Second-line Treatment for Nocturia in Men With LUTS: a Pilot Study
Brief Title: Alpha-blocker Plus Diuretic Combination Therapy as Second-line Treatment for Nocturia in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Seung Paick/M.D.,Ph.D., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mccho
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Nocturia
Keywords: nocturia; bladder; urination disorders; hydrochlorothiazide; terazosin
MeSH Terms: conditions — Nocturia; Urination Disorders | interventions — Hydrochlorothiazide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: combination therapy of terazosin and hydrochlorothiazide

INTERVENTIONS:
Drug: combination therapy of terazosin and hydrochlorothiazide — 25 mg of hydrochlorothiazide eight hours before bedtime and 4 mg of terazosin at bedtime for 4 weeks

SUMMARY:
The aim of the present study was to determine whether the combined administration of a diuretic agent, hydrochlorothiazide, at night would improve the frequency of nocturia unresponsive to alpha-blocker monotherapy in men with LUTS.

DETAILED DESCRIPTION:
Because nocturia may result in sleep disturbances, daytime fatigue, a lower level of general well-being, and an increased risk of falling at night, it is among the most bothersome of the lower urinary tract symptoms (LUTS). Nocturia is related to a variety of conditions such as aging, overactive bladder (OAB), benign prostatic hyperplasia (BPH)/LUTS, medications, diabetes mellitus, diabetes insipidus, anorexia nervosa, and sleep disturbance. In a previous study, we suggested that treatment with terazosin can reduce episodes of nocturia, both subjectively and objectively, in some men with LUTS. Other study showed that in men with nocturnal polyuria, furosemide resulted in a significant reduction in night-time frequency and percentage of the voided volume.

ELIGIBILITY:
Inclusion Criteria:

* no response or < 25% reduction in subjective nocturia by the IPSS question 7 after 4-weeks of treatment with terazosin
* no response or < 25% reduction in objective nocturia by the FVC after 4-weeks of treatment with terazosin
* nocturia on average two times or more per night (according to the FVC) after 4-weeks of terazosin therapy

Exclusion Criteria:

* use of medications for the control of bladder symptoms
* use of sedatives or tranquillisers for treating sleep disturbances
* bladder tumours
* bladder stones
* urethral strictures
* neurogenic bladder dysfunction
* restricted mobility
* working primarily at night
* a documented history or clinical symptoms of prostatitis, prostate cancer, or prostatic intraepithelial neoplasia on biopsy
* serum PSA levels of >20 ng/mL
* a history of prostate surgery or radiotherapy, acute urinary retention or an indwelling catheter
* evidence of acute urinary infection (pyuria and bacteriuria)on urine analysis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
3-day frequency-volume chart | at baseline and at the end of the 4-week therapy

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) question 7 | at baseline and at the end of the 4-week therapy

CONTACTS AND LOCATIONS:
Overall Officials: Min Chul Cho, M.D. Master, Principal Investigator — Department of Urology, Seoul National University College of Medicine
Locations (1):
- Department of Urology, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Result] Cho MC, Ku JH, Paick JS. Alpha-blocker plus diuretic combination therapy as second-line treatment for nocturia in men with LUTS: a pilot study. Urology. 2009 Mar;73(3):549-53; discussion 554-5. doi: 10.1016/j.urology.2008.08.517. Epub 2008 Dec 18. PMID 19100605